CLINICAL TRIAL: NCT01544049
Title: Patients Salpingectomy as a Method of Ovarian Cancer Prevention: A Descriptive Study
Brief Title: Fallopian Tube Removal as a Method of Ovarian Cancer Prevention: A Descriptive Study
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Elizabeth Swisher, Professor, University of Washington
Other Study IDs: STUDY00000276
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Ovarian Cancer
Keywords: fallopian tube removal; salpingectomy; ovarian cancer prevention
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fallopian tube removal: Women who have had one or both fallopian tube(s) removed as method of ovarian cancer prevention.

SUMMARY:
The purpose of this study is to better understand why women choose to have their fallopian tubes removed as a method for ovarian cancer prevention. This will be done through a paper questionnaire and phone interviews. The investigators hope to gain information that will allow us to better counsel women about ovarian cancer prevention.

DETAILED DESCRIPTION:
Women will be found eligible for this study after an eligibility questionnaire given over the phone. If one is found eligible, she will be sent a consent and paper survey to fill out and send back to the research coordinator. Once that is completed, she will be given a phone interview in order answer additional questions of interest. Lastly, the study participant will be contacted once a year over the phone to obtain follow-up information.

ELIGIBILITY:
Inclusion Criteria:

* Female of at least 18 years of age
* Must speak English fluently
* Have had fallopian tubes removed as a method of ovarian cancer prevention

Exclusion Criteria:

* Males
* Females under the age of 18

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who have had their fallopian tubes removed as a method of ovarian cancer prevention.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-12; Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Describe subject experience in undergoing Salpingectomy as a means of riks reduction | At conclusion of study
  Subjects will provide information on their reason for choosing salpingectomy and the process they went through in undergoing this procedure

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Swisher, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States